CLINICAL TRIAL: NCT07379853
Title: Interactive E-Learning for Therapist Training in Exposure Therapy
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Bradley Hospital (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: R41MH139194 (NIH); R41MH139194 (NIH)
Record Dates: First submitted 2026-01-22; First posted 2026-02-02 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-01

CONDITIONS: Therapist Training; ANXIETY DISORDERS (or Anxiety and Phobic Neuroses)
Keywords: Therapist training; Exposure therapy; Anxiety Disorders
MeSH Terms: conditions — Anxiety Disorders; Phobic Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Open Training Trial (Experimental): Therapist will complete the entire eLearning training program
  Interventions: Other: Therapist Training

INTERVENTIONS:
Other: Therapist Training — Therapist training in Exposure Therapy delivery using an eLearning platform

SUMMARY:
The project involves the development of an eLearning platform to train therapists in the delivery of exposure therapy for clients with anxiety disorders and OCD. Following initial development, clinician end users will complete rounds of iterative feedback to inform final development, at which point, therapists will be recruited to complete the entire training program in an open trial.

DETAILED DESCRIPTION:
Despite the existence of numerous well-established evidence-based practices (EBPs) for mental disorders, it has been difficult to disseminate these practices in community settings. Exposure therapy for anxiety disorders represents one of the most glaring examples of this research-to- practice gap. Many practicing therapists have never had the opportunity to receive training in exposure therapy and cite this as a primary barrier to its delivery. To address this gap, investigators need to rethink the way in which they train providers. Recent advances in e-learning offer an exciting opportunity to automate both the didactic and interactive components of these evidence-based training modules-an approach that has potential to vastly improve scalability, thus addressing a primary barrier to accessing the most potent treatment available for anxiety. In this project, the team will develop and initially test an automated eLearning approach for therapists learning exposure therapy. The investigators will leverage evidence-based training content and strategies from their prior work, as well as recent advances in eLearning (e.g., adaptive eLearning). The proposed Phase I STTR study will take place in three stages. Stage one (Development) is a nine-month development period during which PARC Innovations will build an alpha version of the training program in accordance with specifications from the research team and early input from a Multi-perspective Advisory Panel (MAP). The MAP (N=8) will consist of professionals with expertise in commercialization, education & e-learning, and/or technology. In Stage two (End- User Feedback and Optimization), a group of clinician end-users (N = 8) will interact with the platform and provide quantitative and qualitative feedback that will be synthesized by the research team into action items for further development. In stage three (Training Trial), therapists (N=40) will complete 8 hours of e-learning training (self-paced) over three weeks. Usability and training outcomes (e.g., therapist knowledge, self-efficacy) from this pilot trial will support a Phase II STTR project aimed at building out and broadly disseminating this eLearning approach.

ELIGIBILITY:
Inclusion Criteria:

* A practicing therapist providing psychotherapy
* Providing treatment for clients with anxiety conditions

Exclusion Criteria:

- Not employed as a mental health provider

Ages: 21 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Estimated)
Dates: Start 2025-04-17 (Actual); Primary Completion 2027-03-31 (Estimated); Study Completion 2027-03-31 (Estimated)

PRIMARY OUTCOMES:
Therapist Beliefs about Exposure (TBES) | Immediately before initiating the training program and immediately after completing the 10-hour training intervention.
  The TBES is a well-validated, 21-item likert measure of therapist reservations about exposure therapy delivery. Total scores range from 0-84 with higher scores representing more reservations about using exposure therapy with clients.
System Usability Scale (SUS) | Immediately before starting the training program and immediately after completing the 10-hour training intervention
  The SUS is a well-validated measure of usability and acceptability of new innovations. This measure is especially common in the evaluation of new software systems. The measure consists of a 10-item measure on a 5-point likert scale. The scale is converted to a 0-100 score with higher scores indicating higher levels of perceived usability.

CONTACTS AND LOCATIONS:
Locations (1):
- Bradley Hospital, Riverside, Rhode Island, United States

IPD SHARING:
Plan to Share IPD: No